CLINICAL TRIAL: NCT03206905
Title: Safety, Tolerability and Sustained Weight Loss of Immediate Endoscopic Sleeve Gastroplasty (ESG) With Diet Modification and Exercise vs. Early Diet Modification and Exercise and Delayed ESG for the Treatment of Obesity
Brief Title: Safety, Tolerability, and Sustained Weight Loss of Endoscopic Sleeve Gastroplasty With Diet Modification and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1501015803
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Sleeve Gastroplasty (Experimental)
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty; Behavioral: Diet and Exercise
- Diet and exercise only. (Active Comparator)
  Interventions: Behavioral: Diet and Exercise

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty — endoscopic, rather than surgical approach, to perform sleeve gastroplasty
  Arms: Endoscopic Sleeve Gastroplasty
Behavioral: Diet and Exercise — nutritional/exercise counseling

SUMMARY:
The purpose of this study is to compare the effect of endoscopic sleeve gastroplasty (ESG) with diet and exercise, to diet and exercise alone, to see which is better in weight loss reduction. Investigators will also compare the effects of ESG to diet and exercise comorbidities such as diabetes, sleep apnea and high cholesterol as well as the various obesity related hormones.

DETAILED DESCRIPTION:
This is a single center, prospective randomized case control study with an additional non randomized case arm. This study includes two research interventional groups. Groups A: ESG with diet and exercise modules. Group B: Diet and exercise modules only. Investigators propose to compare ESG to behavioral modification including diet and exercise for patients who have a BMI greater than or equal to 40 kg/m2 or greater than or equal to 30 kg/m2 with 1 or more obesity related co-morbidity and who cannot undergo conventional bariatric surgery(or decline the surgical option). Investigators will also compare the effects of ESG to diet and exercise on comorbidities such as diabetes, sleep apnea and high cholesterol as well as the various obesity related hormones.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 40 kg/m2, greater than or equal to to 30 kg/m2 with 1 more obesity related co-morbidity, or or greater than or equal to 35 kg/m2 without co-morbidity

Co-morbidities include:

1. Sleep apnea (STOP-BANG questionnaire and polysomnography)
2. BP >130/80 or on hypertension meds.
3. A1c > or = to 5.7, fasting >100 OR RANDOM >126, exclude 6.5 and above
4. Waist circumference >102, or 40 inches if male or >80 cm 35 inches if female
5. Metabolic syndrome (3 criteria, blood pressure, waist circumference, triglycerides > 150 or HDL < 50/40)

   * Failure to respond to non-invasive weight loss management for at least 6 months.
   * Valid health insurance to cover the cost of procedure and standard of care pre-and post-procedure management/workup.

Exclusion Criteria:

* Untreated endocrine diseases (diabetes, thyroid disorder, pituitary disorder, and sex gland disorder).
* diabetes or A1c >6.5
* Heart Disease, for example, arrhythmia, heart failure, myocardial infarction.
* Kidney disease with serum creatinine greater than 2.5 mg/dl.
* Cerebrovascular disease, for example, stroke or otherwise unable to exercise.
* Any pregnant or lactating women or who have had childbirth within 6 months.
* Any patients on retinoid therapy or undergoing retinoid therapy that will not last throughout the length of the trial.
* Patients with significant psychiatric disorder.
* Any other chronic condition deemed unsuitable to undergo either arm of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Percentage of Total Body Weight Loss | 6 months
  To compare mean percentage weight loss achieved via ESG with diet modification and exercise, vs. diet modification and exercise only in patients who cannot undergo conventional bariatric surgery for obesity (with BMI greater than or equal to 40 kg/m2 or greater than or equal to 30 kg/m2 with 1 or more obesity related co-morbidity).

CONTACTS AND LOCATIONS:
Overall Officials: Reem Sharaiha, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Weill Cornell Medicine, Division of Gastroenterology & Hepatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided